CLINICAL TRIAL: NCT05651412
Title: Normative Data of Dynamic Gait Index and 5 Time Sit to Stand Test Among Elderly Population and Correlation With Anthropometric Parameters
Brief Title: Normative Data of Dynamic Gait Index and 5 Time Sit to Stand Test Among Elderly Population
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: Semera
Record Dates: First submitted 2022-10-21; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Fall; Old Age; Debility
Keywords: Anthropometrics; DGI; Five time sit to stand test
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dynamic gait index and 5 time sit to stand test — dynamic gait index and 5 time sit to stand test was administered to all sample size of 400

SUMMARY:
The goal of this observational study is to measure the normative data for dynamic gait index and 5 time sit to stand test in elderly population. This study aimed for to take normative measurement of dynamic gait index and five time sit to stand test among elderly population and to compare the preliminary values of above mentioned tests with age.

DETAILED DESCRIPTION:
Anthropometric factors affect the stability limits of the individual and can affect the motor strategies relating to balance control. The core elements of anthropometry are height, weight, body mass index (BMI), body circumferences (waist, hip, and limbs), and skin-fold thickness. Some anthropometric variables, such as body mass, are directly related to postural balance. Due to lack of normative data for dynamic gait index and five times sit to stand test in elderly population, this study aimed to formulate normative values for dynamic gait index and five times sit to stand test among elderly and correlation with anthropometric measures. Objectives: The objective of this study was to take normative measurement of dynamic gait index and five times sit to stand test among elderly population and to compare the preliminary values of above mentioned tests with age. All possible elder population was taken in current study to calculate the normative values of these two tests, five times STS to measure the ability to get up from a chair and DGI to record dynamic gait tasks in elder people

ELIGIBILITY:
Inclusion Criteria:

* 45-60 years elderly population.
* Both male and female were included in given age group.
* Older adults ambulate without a device or assistance.
* Population who has no deformity will be included.

Exclusion Criteria:

* Older adults who cannot ambulate were excluded
* Pregnant females were excluded from this study
* Population having any deformities was not included in this study.
* Any participants suffering from malignancy, infection or taking anticoagulant therapy were also excluded.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Data was collected from old age home in Lahore. Sample size of 400 subjects was chosen.
  Group 1: 45-50 years Group 2: 50-55 years Group 3: 55-60 years
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait index | 8 weeks
  8 functional walking tests are performed by the subject and marked out of three according to the lowest category which applies. 24 is the total individual score possible. Scores of 19 or less have been related to increase incidence of falls.
  Equipment needed
  Box (Shoebox), Cones (2), Stairs, 20' walkway, 15" wide
  Completion Time
  15 minutes
5 times sit to stand test | 8 weeks
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and identify movement strategies a patient uses to complete transitional movements.
  The equipment need in performing 5XSST test includes: Stopwatch and chair with straight back (43-45 cm, 17-18 inches high). Then the instruction is given by asking the test taker to sit on the chair by resting their back. Also, the test taker is instructed to fold their arms across their chest. Then the test taker should be instructed to do sit-to-stand five times, as quickly as possible, at the count of go and without their back or leg resting on the chair between the interval of repetition

CONTACTS AND LOCATIONS:
Overall Officials: Sumera Azam, MS, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Maria Idrees, Lahore, Punjab Province
  - Riphah International University, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No